CLINICAL TRIAL: NCT05378087
Title: Non-randomized Concurrent Controlled Trial of Surgery Staging or Image Staging of Locally Advanced Cervical Cancer
Brief Title: Comparing the Efficacy of Surgery Staging and Image Staging of Locally Advanced Cervical Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Dongling Zou, Director of Gynecologic Oncology Department, Chongqing University Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQGOG0106
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Locally Advanced Cervical Cancer
Keywords: surgery staging; image staging; Locally advanced cervical cancer; PFS

STUDY DESIGN:
Intervention Model Description: This is a non-randomized controlled concurrent trial. According to the patients' voluntary choice, they are enrolled on the surgery staging group or image staging group. All patients are evaluated by CT(≥32 slices) or MRI(≥1.5T) or PET/CT. The criteria for positive pelvic or para-aortic lymph nodes (one of the following): ① CT or MRI show more than one positive lymph node with a short diameter ≥ 15mm; ② PET/CT shows more than one positive lymph node with SUV ≥ 2.5; ③ If CT or MRI show positive lymph node with a short diameter between 10mm and 15mm, PET / CT should further verify that it is a positive lymph node with SUV ≥ 2.5.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Image staging group (Active Comparator): Standard chemoradiation (Pelvic EBRT/Extended-field EBRT + concurrent platinum-containing chemotherapy + brachytherapy).
  Interventions: Radiation: Concurrent chemoradiation
- Surgery staging group (Experimental): Open/minimally invasive para-aortic lymph node dissection followed by chemoradiation (Pelvic EBRT/Extended-field EBRT + concurrent platinum-containing chemotherapy + brachytherapy).
  Interventions: Procedure: Open/minimally invasive para-aortic lymph node dissection followed by concurrent chemoradiation

INTERVENTIONS:
Radiation: Concurrent chemoradiation — Standard concurrent chemoradiation: A point/HCR-CTV D90 ≥80Gy (+20%) by using IMRT or TOMO technics. Patients with image-positive common iliac lymph nodes or para-aortic lymph nodes receive extended-field EBRT. Brachytherapy should begin after 15-20F external radiotherapy. A radiation dose for the image-positive nodes can range from 55Gy to 60Gy. Five cycles of concurrent platinum-containing chemotherapy (Cisplatin 40mg/m2 q1w or Carboplatin AUC=2 q1w, Window period one week) and CCRT should be completed within 56 days. CCRT one week later, if the cervix biopsy shows residual tumour and/or imaging (CT/MRI/PET/CT) indicates that there are still positive lymph nodes in the pelvic and abdominal cavity, three cycles of adjuvant chemotherapy (TP: Paclitaxel 135mg/m2, Cisplatin 50mg/m2, q3w or TC: Paclitaxel 135mg/m2, Carboplatin AUC=4, q3W; Window period 2 weeks) ± brachytherapy will be performed (A point/HR-CTV D90 ≤ 96Gy).
  Arms: Image staging group
Procedure: Open/minimally invasive para-aortic lymph node dissection followed by concurrent chemoradiation — Open/minimally invasive para-aortic lymph node dissection followed by concurrent chemoradiation. (height of lymph node dissection: At least the inferior mesenteric artery. Chemoradiation should be performed postoperatively within 28 days.) The chemoradiation is consistent with the image staging group, except for extended-field EBRT determined by pathological positive para-aortic lymph nodes.
  Arms: Surgery staging group

SUMMARY:
The study is a domestic multicenter, prospective, non-randomized controlled concurrent trial. It will be assessed whether surgery staging on locally advanced cervical cancer is superior to image staging for improving progression-free survival and overall survival.

DETAILED DESCRIPTION:
All eligible patients will be divided into the following two treatment groups nonrandomly.

Image staging group: standard chemoradiation (Pelvic EBRT/Extended-field EBRT + concurrent platinum-containing chemotherapy+brachytherapy).

Surgery staging group: open/minimally invasive para-aortic lymph node dissection followed by concurrent chemoradiation. (Level of lymph node dissection: At least the inferior mesenteric artery. Chemoradiation will be conducted within 28 days postoperatively.)

ELIGIBILITY:
Inclusion Criteria:

1. The patients with good compliance, voluntarily signed the informed consent form and participated in the study.
2. Histopathology: squamous cell carcinoma, adenocarcinoma, adenosquamous cell carcinoma
3. Stage (FIGO2018): IB3, IIA2, IIB-IVA;
4. ECOG score: 0 ~ 1;
5. The expected survival >6 months;
6. The result of a pregnancy test (serum or urine) within seven days must be negative for women of childbearing age, who must take contraception during the trial.

Exclusion Criteria:

1. Activity or uncontrol severe infection;
2. Liver cirrhosis or other decompensated liver disease;
3. A history of immune deficiency, including HIV positive or a congenital immunodeficiency disease;
4. Chronic renal insufficiency or renal failure;
5. Other malignancies were diagnosed within five years or needed treatments;
6. Myocardial infarction, severe arrhythmia and congestive heart failure with grade ≥2 (New York heart association);
7. The CT/MRI/PET/CT show that the para-aortic lymph nodes are positive;
8. A history of pelvic artery embolization;
9. A history of pelvic radiotherapy;
10. A history of partial hysterectomy or radical hysterectomy;
11. A history of severe allergic reaction to platinum drugs;
12. The drugs for the treatment of concomitant disease seriously impaired liver or kidney function, such as tuberculosis;
13. Patients who cannot understand the research regimen and refuse to sign the informed consent form;
14. Other concomitant diseases or special conditions seriously endanger the patient's health or interfere with the trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1956 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 3 years
  Progression-free survival

SECONDARY OUTCOMES:
OS | 3 years and 5 years
  3-year and 5-year Overall Survival
Complication | 1 year
  Some conditions caused by surgery or chemoradiation.

CONTACTS AND LOCATIONS:
Overall Officials: Dongling Zou, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The study involves confidentiality and patients' privacy protection.

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Bhatla N, Berek JS, Cuello Fredes M, Denny LA, Grenman S, Karunaratne K, Kehoe ST, Konishi I, Olawaiye AB, Prat J, Sankaranarayanan R, Brierley J, Mutch D, Querleu D, Cibula D, Quinn M, Botha H, Sigurd L, Rice L, Ryu HS, Ngan H, Maenpaa J, Andrijono A, Purwoto G, Maheshwari A, Bafna UD, Plante M, Natarajan J. Revised FIGO staging for carcinoma of the cervix uteri. Int J Gynaecol Obstet. 2019 Apr;145(1):129-135. doi: 10.1002/ijgo.12749. Epub 2019 Jan 17. PMID 30656645
- [Background] Martinez A, Angeles MA, Querleu D, Ferron G, Pomel C. How should we stage and tailor treatment strategy in locally advanced cervical cancer? Imaging versus para-aortic surgical staging. Int J Gynecol Cancer. 2020 Sep;30(9):1434-1443. doi: 10.1136/ijgc-2020-001351. Epub 2020 Aug 11. PMID 32788263
- [Background] Choi HJ, Ju W, Myung SK, Kim Y. Diagnostic performance of computer tomography, magnetic resonance imaging, and positron emission tomography or positron emission tomography/computer tomography for detection of metastatic lymph nodes in patients with cervical cancer: meta-analysis. Cancer Sci. 2010 Jun;101(6):1471-9. doi: 10.1111/j.1349-7006.2010.01532.x. Epub 2010 Feb 11. PMID 20298252
- [Background] Kang S, Kim SK, Chung DC, Seo SS, Kim JY, Nam BH, Park SY. Diagnostic value of (18)F-FDG PET for evaluation of paraaortic nodal metastasis in patients with cervical carcinoma: a metaanalysis. J Nucl Med. 2010 Mar;51(3):360-7. doi: 10.2967/jnumed.109.066217. Epub 2010 Feb 11. PMID 20150275
- [Background] Gouy S, Seebacher V, Chargari C, Terroir M, Grimaldi S, Ilenko A, Maulard A, Genestie C, Leary A, Pautier P, Morice P, Deandreis D. False negative rate at 18F-FDG PET/CT in para-aortic lymphnode involvement in patients with locally advanced cervical cancer: impact of PET technology. BMC Cancer. 2021 Feb 6;21(1):135. doi: 10.1186/s12885-021-07821-9. PMID 33549033
- [Background] Gouy S, Morice P, Narducci F, Uzan C, Martinez A, Rey A, Bentivegna E, Pautier P, Deandreis D, Querleu D, Haie-Meder C, Leblanc E. Prospective multicenter study evaluating the survival of patients with locally advanced cervical cancer undergoing laparoscopic para-aortic lymphadenectomy before chemoradiotherapy in the era of positron emission tomography imaging. J Clin Oncol. 2013 Aug 20;31(24):3026-33. doi: 10.1200/JCO.2012.47.3520. Epub 2013 Jul 15. PMID 23857967
- [Background] Gouy S, Morice P, Narducci F, Uzan C, Gilmore J, Kolesnikov-Gauthier H, Querleu D, Haie-Meder C, Leblanc E. Nodal-staging surgery for locally advanced cervical cancer in the era of PET. Lancet Oncol. 2012 May;13(5):e212-20. doi: 10.1016/S1470-2045(12)70011-6. PMID 22554549
- [Background] Gold MA, Tian C, Whitney CW, Rose PG, Lanciano R. Surgical versus radiographic determination of para-aortic lymph node metastases before chemoradiation for locally advanced cervical carcinoma: a Gynecologic Oncology Group Study. Cancer. 2008 May 1;112(9):1954-63. doi: 10.1002/cncr.23400. PMID 18338811
- [Background] Frumovitz M, Querleu D, Gil-Moreno A, Morice P, Jhingran A, Munsell MF, Macapinlac HA, Leblanc E, Martinez A, Ramirez PT. Lymphadenectomy in locally advanced cervical cancer study (LiLACS): Phase III clinical trial comparing surgical with radiologic staging in patients with stages IB2-IVA cervical cancer. J Minim Invasive Gynecol. 2014 Jan-Feb;21(1):3-8. doi: 10.1016/j.jmig.2013.07.007. Epub 2013 Jul 31. PMID 23911560
- [Background] Kohler C, Mustea A, Marnitz S, Schneider A, Chiantera V, Ulrich U, Scharf JP, Martus P, Vieira MA, Tsunoda A. Perioperative morbidity and rate of upstaging after laparoscopic staging for patients with locally advanced cervical cancer: results of a prospective randomized trial. Am J Obstet Gynecol. 2015 Oct;213(4):503.e1-7. doi: 10.1016/j.ajog.2015.05.026. Epub 2015 May 15. PMID 25986030
- [Background] Lai CH, Huang KG, Hong JH, Lee CL, Chou HH, Chang TC, Hsueh S, Huang HJ, Ng KK, Tsai CS. Randomized trial of surgical staging (extraperitoneal or laparoscopic) versus clinical staging in locally advanced cervical cancer. Gynecol Oncol. 2003 Apr;89(1):160-7. doi: 10.1016/s0090-8258(03)00064-7. PMID 12694671